CLINICAL TRIAL: NCT00954915
Title: A Phase 2a, Open Label, Multiple-Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Teplizumab in Adults With Moderate or More Severe Psoriasis
Brief Title: Safety Study of the Monoclonal Antibody Teplizumab (MGA031) in Subjects With Moderate or More Severe Psoriasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Injection site reaction met protocol-defined stopping criteria.
Sponsor: MacroGenics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA031-04
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis
Keywords: chronic plaque psoriasis; psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — teplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- teplizumab (Experimental): Anti CD-3 monoclonal antibody
  Interventions: Biological: teplizumab

INTERVENTIONS:
Biological: teplizumab — Cohorts 1-5: escalating doses of subcutaneously administered teplizumab; cohort 6: intravenous administration of maximum tolerated subcutaneous dose.
  Other Names: MGA031

SUMMARY:
The purpose of this study is to determine whether teplizumab is safe when administered subcutaneously (by needle under the skin) in subjects with psoriasis. The study will also evaluate how long teplizumab stays in the blood and how long it takes for it to leave the body, what is the highest dose that can safely be given, and whether it improves psoriasis.

DETAILED DESCRIPTION:
This study will test the hypotheses that therapeutic modulation of T-cell function by teplizumab is well tolerated in subjects with moderate or more severe psoriasis, and that this treatment ameliorates the immunopathology of psoriasis. This study will evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of subcutaneous (SC) administration for 6 days. Once the SC maximum tolerated dose is identified, this dose will be administered to a cohort of subject by intravenous for comparison of PK and PD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis that has been present for more than 6 months and involves at least 10% Body Surface Area (BSA).
* Baseline LS-PGA score of moderate or greater severity.
* Weight <= 125 kg (276 lb) and a BSA <= 2.5 m^2.

Exclusion Criteria:

* Clinically significant flare of psoriasis during the 12 weeks before enrollment.
* Guttate, erythrodermic, palmoplantar, or pustular (von Zumbusch) psoriasis
* Orally administered systemic psoriasis therapy or phototherapy within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks before enrollment.
* Prior administration of a biologic agent/monoclonal antibody within 12 weeks before enrollment or 5 half-lives of the agent, whichever is greater.
* Prior otelixizumab, OKT®3, or teplizumab.
* Treatment within the last 30 days with a non-biologic drug or device that has not received regulatory approval for any indication at the time of study entry or are unwilling to forgo experimental treatment other than teplizumab during this study.
* Treatment with live vaccine within 8 weeks before enrollment or during study; vaccination with an antigen or killed organism during the study, within 8 weeks before enrollment, or 8 weeks after dosing.
* Evidence of active infection.
* Positive IgM test for hepatitis A.
* History of or positive test for hepatitis B, C, or D.
* History of or positive test for HIV.
* Are immunocompromised, have had recent or current serious systemic or local infection, clinical or radiological evidence of active tuberculosis, or evidence of latent TB infection.
* History of chronic liver disease, peripheral vascular disease, cerebrovascular disease, cardiovascular disease, or epilepsy.
* Current serious or unstable illnesses or allergies.
* Clinically significant laboratory abnormalities.
* Presence of serological reactivity to teplizumab (in subjects previously treated with therapeutic antibodies).
* Clinically significant ECG abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began at two academic institutions in April 2010 and was halted on December 17, 2010 after the first subject had an injection site reaction that met study stopping criteria.
Period: Overall Study
Arm/Group | Teplizumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Teplizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AE)
Description: Primary endpoints include safety data such as vital signs, physical examinations, electrocardiograms, AE reports, and laboratory test results.
Time Frame: Day 0 through Day 84
Population: One subject was enrolled and followed per protocol. This subject's data are described in the adverse events summary.
Measure: Number; unit: Participants
Groups:
- Teplizumab: anti-CD3 monoclonal antibody
Arm/Group | Teplizumab
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Participants Improved on Lattice System Physician's Global Assessment (LS-PGA)
Description: The LS-PGA score is determined by estimating the extent of body surface area involved by psoriasis and rating plaque qualities (elevation, erythema, scaling) averaged over the entire body. LS-PGA score is then determined using available software. LS-PGA ranks involvement on an 8 point scale from clear, almost clear, mild, mild to moderate, moderate, moderate to severe, severe, and very severe. Participants who have an improvement of one or more steps in the LS-PGA will be considered to have met the primary criteria for a clinical response.
Time Frame: Day 0, 14, 28, 63 and 84
Population: Data were not collected due to early termination of the study.
Arm/Group | Teplizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Improved on the Psoriasis Area and Severity Index (PASI)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of plaque scale, erythema, and plaque induration (thickness) in each region, yielding an overall score of 0 for no psoriasis to a maximum of 72 for severe disease.
Time Frame: Day 0, 14, 28, 63 and 84
Population: Data were not collected due to early termination of the study.
Arm/Group | Teplizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Physician's Global Assessment (PGA)
Description: The PGA rates the subject's psoriasis relative to baseline as 1 (100% clearing), 2 (excellent: 75% through 99% clearing with striking improvement), 3 (good: 50% through 74% clearing with moderate improvement), 4 (fair: 25% through 49% clearing with slight improvement), 5 (poor: 0% through 24% clearing with little or no change), or 6 (worsening). Involvement of body-surface area, induration, scaling, and erythema are taken into account.
Time Frame: Day 0, 14, 28, 63 and 84
Population: Data were not collected due to early termination of the study.
Arm/Group | Teplizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Teplizumab Blood Levels
Time Frame: Day 0 through Day 84
Population: Data were not collected due to early termination of the study.
Arm/Group | Teplizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Teplizumab
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teplizumab (N=1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Injection site reaction condition aggravated (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
CD3 lymphocytes decreased (Investigations) | 1 (1)
Platelet count increased (Blood and lymphatic system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated, with only 1 subject enrolled, due to meeting the study criteria for discontinuation regarding local or regional injection site reactions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days